CLINICAL TRIAL: NCT06461208
Title: PROMISE Trial: A PROspective Randomised Double-blind Parallel Group Placebo-controlled Multicentre Trial of Faecal MIcrobiota tranSplantation to Improve the Primary outcomE (First Hospitalisation Due to Infection) in Patients With Cirrhosis Over 24 Months
Brief Title: A PROspective Faecal MIcrobiota tranSplantation Trial to Improve outcomEs in Patients With Cirrhosis
Acronym: PROMISE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: St George's, University of London (Other); Guy's and St Thomas' NHS Foundation Trust (Other); Imperial College London (Other); King's College Hospital NHS Trust (Other); BRITISH LIVER TRUST (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1004822; 2022-000300-35 (EudraCT Number); NIHREME130730 (Other Grant/Funding Number: NIHR EME); ISRCTN17863382 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2024-06-04; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-05

CONDITIONS: Liver Cirrhosis
Keywords: Fatty Liver Alcoholic; Alcohol-related Liver Disease; Metabolic dysfunction-Associated Steatotic Liver Disease; Liver Cirrhosis; MASLD; MASLD-ALD overlap cirrhosis; ALD; Faecal Microbiota Transplant; Metabolic Fatty Liver Disease; Fatty Liver Disease; Gut Microbiota; Cirrhosis; PROMISE
MeSH Terms: conditions — Liver Cirrhosis; Fatty Liver, Alcoholic; Non-alcoholic Fatty Liver Disease; Fibrosis

STUDY DESIGN:
Intervention Model Description: Patients will be randomised 1:1 to FMT or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants, Chief Investigator, Site Principal Investigators and outcome assessors will be fully blinded throughout the trial. The site pharmacy trials team and the nurse administering the treatment will be unblinded to a patients treatment allocation.
  The senior statistician will also be fully blinded, but the junior statistician will be unblinded from the 1st DMC meeting with data onwards.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Encapsulated FMT (Experimental)
  Interventions: Drug: Encapsulated FMT
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Encapsulated FMT — Encapsulated Faecal Microbiota Transplant
  Arms: Encapsulated FMT
Other: Placebo — The placebo product contains microcrystalline methylcellulose. It is supplied as a size 0, Swedish Orange Delayed-Release capsule (DRCap) and provides a complete match with regards to the appearance (e.g., dimensions, colour) to the FMT capsules.
  Arms: Placebo

SUMMARY:
A feasibility trial called PROFIT has previously shown that FMT administered endoscopically into the jejunum in patients with cirrhosis is safe and feasible and have identified some potential mechanisms of action that warrant further interrogation. The aim of the PROMISE Trial is to evaluate the efficacy and mechanisms of action of encapsulated FMT (versus placebo) to reduce infection and mortality in patients with alcohol-related and metabolic dysfunction-Associated Steatotic Liver (MASLD) cirrhosis.

DETAILED DESCRIPTION:
There is an evolving crisis of chronic liver disease (CLD) in the UK and it is the only major chronic disease which is on the rise. The advanced stages of CLD, known as cirrhosis (a hardening and scarring of the liver), is the third biggest cause of death and loss of working life years behind heart disease and self-harm. People die from cirrhosis young with more than 1 in 10 in their 40s.

Patients with cirrhosis are very susceptible to infections, antibiotics become ineffective and patients may become infected with 'super bugs'. There is an urgent need for antibiotic-free approaches. The body contains trillions of microscopic organisms called bacteria which play an important role in keeping us healthy. Many of these bacteria live within our bowel and help our immune system fight infection. There are increased numbers of 'unfriendly' bowel bacteria in patients with cirrhosis which emit substances that are harmful to health and disrupt the immune system.

It could be beneficial to replace the unfriendly bowel bacteria in patients with cirrhosis with bacteria donated from a healthy person by performing a type of bowel bacteria transplant (known as faecal microbiota transplantation or FMT). The PROFIT trial was recently performed as a preliminary trial of FMT which was placed into the bowel with the help of a flexible camera (endoscopy). The study showed FMT was safe with no serious side effects, but patients told us they would prefer to take tablets rather than have an endoscopy. The chief investigator and her team have therefore made a capsule which contains dried stool from a healthy donor. Participants will need to take 5 of these capsules to achieve the same dose.

The PROMISE clinical trial is to test whether treating patients with FMT capsules will reduce the likelihood of them getting an infection by measuring the time it takes to develop an infection resulting in hospital admission. This will be compared to a 'dummy' capsule that contains no FMT (placebo). Patients will be selected at random to have FMT treatment or placebo and both the study team and the patients will not know which treatment they are taking. Participants will need to take 5 capsules every 3-months. Participants will continue treatment for a total of 21-months or until they develop their first infection leading to hospital admission and will be followed-up for a maximum of 2-years.

This study will also examine if having FMT will reduce the side effects of cirrhosis and if it has beneficial effects on the liver and immune system. The investigator team will study whether it reduces hospital admissions, the incidence of 'super-bug' infections and death. Laboratory studies will look at whether FMT treatment will help the immune system fight infection.

The World Health Organisation describes the resistance of bacteria to the effects of antibiotics as one of the biggest threats to global health. The discovery of new antibiotics has not kept pace. The government's white paper proposes a 5-year plan to tackle resistance to antibiotics. Consultation with our patient co-applicant, patient advisory group, The British Liver Trust and Guts UK Charity have highlighted recurrent hospitalisation, over-use of antibiotics and fear of acquiring a 'super-bug' as being important priorities to patients. The results and study findings will be published in conjunction with patient support groups, the wider media and the NHS. The investigator will ensure the research impacts on the management of patients with CLD and shapes policy and guideline development.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years
2. Confirmed Alcohol-related (ALD) or Metabolic dysfunction-Associated Steatotic Liver Disease (MASLD) or MASLD-ALD Overlap cirrhosis based on clinical, radiological and/or histological criteria.
3. MELD score 8-16 28
4. Patients with alcohol-related cirrhosis must have been abstinent for a minimum of 4 weeks prior to randomisation.
5. Patients must be deemed to have the capacity to provide written informed consent to participate.

Exclusion Criteria:

1. Severe or life-threatening food allergy (e.g., peanut allergy)
2. Pregnancy or planned pregnancy*. Urine testing will be performed at screening to rule out pregnancy in females.
3. Breast-feeding
4. Patients treated for acute variceal bleeding, infection, overt hepatic encephalopathy, bacterial peritonitis or ACLF within 14 days prior to randomisation.
5. Active alcohol consumption of >20 grams/day [1 unit of alcohol contains 10mLs or 8g of alcohol]
6. Had a previous liver transplant
7. Patients with inflammatory bowel disease.
8. Patients with coeliac disease.
9. Patients with a history of prior gastrointestinal resection or surgery that could change the gut microbiome or result in bacterial overgrowth e.g. gastric bypass
10. Active malignancy including hepatocellular carcinoma
11. Patients with an expected life expectancy <6 months or listed for liver transplantation
12. Infected with HIV, hepatitis B or C [patients who have undetectable hepatitis B or C DNA/RNA can be recruited].
13. Patients who have received antibiotics or probiotics (excluding food stuffs containing 'live bacteria' such as live yoghurts, kefir, fermented vegetables such as sauerkraut/kombucha or cheese) within 7 days prior to randomisation. Protocol Version 3.0 - 03/11/2023 33
14. Swallowing disorder, oral-motor dyscoordination or likely inability/unwillingness to ingest study medication.
15. Patients who have received another investigational drug or device within 4 months prior to randomisation.
16. Patients, who in the opinion of the PI, have a medical condition, or other relevant psychological, familial, or social factor that may jeopardise their health, compliance, or influence the trial integrity in any way.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Defined infection resulting in hospital admission | From date of randomisation until the date of first hospitlisation, assessed up to Month 24.
  To evaluate the efficacy of encapsulated FMT to reduce the susceptibility of infection in patients with cirrhosis measured by the time to first infection resulting in hospitalisation.

SECONDARY OUTCOMES:
Incidence of decompensating events | Screening - End of Visit (Month 24)
  All types of decompensating events will be included:
  i. hepatic encephalopathy, ii. new-onset ascites, iii. variceal bleeding and iv. spontaneous bacterial peritonitis.
Progression to ACLF (Acute on Chronic Liver Failure) i.e. the development of one or more organ failure | Screening - End of Visit (Month 24)
All-cause culture-confirmed infection | Screening - End of Visit (Month 24)
Incidence of antibiotic usage | Screening - End of Visit (Month 24)
Occurrence of AMR (Anti-Microbial Resistance) | Screening - End of Visit (Month 24)
  (including skin and nose colonisation with methicillin-resistant Staphylococcus aureus (MRSA), vancomycin-resistant Enterococci (VRE), extended spectrum beta-lactamase producing bacteria (ESBL), fluoroquinolone-resistant gram negative and linezolid-resistant Enterococci (LRE).
Hospitalisation rates (liver-related and all-cause) (time to event) including the length of stay (time to discharge among hospitalised participants) and admission to high dependency/intensive care. | Screening - End of Visit (Month 24)
Change in liver disease severity scores | Screening - End of Visit (Month 24)
  Child Pugh Score Score range: Min 5 - Max 15 (The higher score, the more worse outcome)
Change in liver disease severity scores | Screening - End of Visit (Month 24)
  MELD Score (Model for End stage Liver Disease) Score range: Min 6 - Max 40 (The higher score, the more worse outcome)
Change in liver disease severity scores | Screening - End of Visit (Month 24)
  UKELD Score (UK for End stage Liver Disease) Score range: Min 40 - Max 80 (The higher score, the more worse outcome)
Change in quality of life (EQ-5D-5L) scores | Screening - End of Visit (Month 24)
  EQ-5D-5L Score (EuroQol-5 Dimension- 5 Levels) Score range: Min 11111 - Max 55555 (The higher score, the more worse outcome)
Change in depression and anxiety scores (using HADS) | Screening - End of Visit (Month 24)
  HADS Score (Hospital Anxiety Depression Scale) Score range: Min 0 - Max 21 (The higher score, the more worse outcome) Data for anxiety and depression to be cateogorised separately.
All-cause mortality and liver-related mortality. | Screening - End of Visit (Month 24)
Change in alcohol use disorder-related events in patients enrolled with alcohol-related cirrhosis as assessed by the alcohol-use disorders identification test (AUDIT score) | Screening - End of Visit (Month 24)
  AUDIT Score (Alcohol Use Disorder Identification Test) Score range: Min 0 - Max 40 (The higher score, the more worse outcome)
Change in urinary ethyl glucuronide/ethyl sulphate levels if tested as part of the standard of care. | Screening - End of Visit (Month 24)

CONTACTS AND LOCATIONS:
Locations (16):
- United Kingdom (16):
  - Royal Bournemouth Hospital, Bournemouth
  - Southmead Hospital, Bristol
  - Bristol Royal Infirmary, Bristol
  - Royal Derby Hospital, Derby
  - Ninewells Hospital, Dundee
  - Queen Elizabeth Hospital, Gateshead
  - Queen Elizabeth University Hospital, Glasgow
  - Hull Royal Infirmary, Hull
  - St. James University Hospital, Leeds
  - King's College Hospital NHS Foundation Trust, London
  - St. George's University Hospital NHS Foundation Trust, London
  - St. Mary's Hospital, London
  - Freeman Hospital, Newcastle upon Tyne
  - Royal Gwent Hospital, Newport
  - Queen's Medical Centre, Nottingham
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: No